CLINICAL TRIAL: NCT02847936
Title: The Effect of Triclosan-coated Sutures for Reducing Risk of Surgical Site Infection After Episiotomy: A Prospective Randomized Controlled Trial
Brief Title: Efficacy of Triclosan-coated Sutures in the Episiotomy
Acronym: EPISIOVIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Amira Ayachi, University Assistant in Obstetrics and gynecology, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: episio1
Record Dates: First submitted 2016-07-22; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Episiotomy
Keywords: triclosan; sutures; infection
MeSH Terms: conditions — Infections | interventions — Polyglactin 910; Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- VICRYL PLUS (Active Comparator): triclosan-coated sutures
  Interventions: Procedure: vicryl plus suture
- VICRYL (Active Comparator): non antibacterial coated sutures
  Interventions: Procedure: vicryl suture

INTERVENTIONS:
Procedure: vicryl plus suture — episiotomy with triclosan-coated sutures
  Arms: VICRYL PLUS
Procedure: vicryl suture — episiotomy with non antibacterial coated suture
  Arms: VICRYL

SUMMARY:
Surgical repair of perineal lesions after delivery can be associated with infection of the surgery site. The aim of this study was to compare the surgical site infection with triclosan-coated suture (Vicryl Plus) versus coated suture (Vicryl) in the episiotomy after delivery.

DETAILED DESCRIPTION:
Women undergoing planned were randomized to either episiotomy suture with VICRYL PLUS or VICRYL. The primary outcome measures were number of sutures used and the development of hematoma, seroma, surgical site infection (SSI) or wound disruption one week after episiotomy. Secondary outcome measures were the cost of the treatment with or without infection, and scar evaluation (wound complication).

Data were analyzed according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who had had an episiotomy at the delivery
* vaginal delivery
* no further perineal or vaginal lesions present

Exclusion Criteria:

* collagen disease
* known immunodeficiency
* Clinical signs of infection at the time of episiotomy
* History of keloids and a medical disorder that could affect wound healing
* Hypersensitivity to any of the suture materials used in the protocol
* Diabetes mellitus
* Disorders requiring chronic corticosteroid use or immunosuppression
* Instrumental extraction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
number of sutures used | two hours
number of patients with wound complications (infection, hematoma, disruption) | one week

SECONDARY OUTCOMES:
cost of the treatment with and without infection | two weeks
  cost of the treatment with and without infection
number of patients with adverse outcomes | two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bougatfa, Bizerte, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guo J, Pan LH, Li YX, Yang XD, Li LQ, Zhang CY, Zhong JH. Efficacy of triclosan-coated sutures for reducing risk of surgical site infection in adults: a meta-analysis of randomized clinical trials. J Surg Res. 2016 Mar;201(1):105-17. doi: 10.1016/j.jss.2015.10.015. Epub 2015 Oct 23. PMID 26850191